CLINICAL TRIAL: NCT03112538
Title: Improving Glycaemic Control in Malaysian Patients With Type 2 Diabetes Mellitus With Insulin Pump Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinical Research Centre, Malaysia (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Nurain Mohd Noor, Consultant Endocrinologist, Clinical Research Centre, Malaysia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NERP14-019
Record Dates: First submitted 2016-10-12; First posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: insulin pump; basal bolus insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Infusion Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin pump (Active Comparator): Medtronic Minimed Paradigm Veo Insulin Pump utilising rapid acting insulin Glulisine or Aspart
  Interventions: Device: Insulin Pump; Drug: Multiple daily injections of insulin
- Multiple daily injections of insulin (Active Comparator): Multiple daily injections consisting of a single basal insulin injection(Glargine) and 3 bolus insulin injections (rapid acting insulin Glulisine or Aspart) before each meal
  Interventions: Device: Insulin Pump; Drug: Multiple daily injections of insulin

INTERVENTIONS:
Device: Insulin Pump — Medtronic Minimed Paradigm Veo Insulin Pump
Drug: Multiple daily injections of insulin — Multiple daily injections which consist of a single injection of basal insulin(insulin Glargine) and 3 injections of bolus insulin(rapid acting insulin Glulisine or Aspart) before each meal
  Other Names: Basal bolus injections of insulin

SUMMARY:
The purpose of this study is to evaluate the comparative efficacy of insulin pump therapy versus multiple daily injections in insulin-taking type 2 diabetes mellitus who are sub-optimally controlled with premixed insulin regimen. This research is necessary because many patients with type 2 diabetes mellitus do not meet their glucose targets.

In advanced Type 2 diabetes mellitus, many patients develop worsening diabetes control and unable to reach the glucose targets despite intensive insulin regimens.This is further complicated by the risks of low blood sugar and weight gain. These limitations of multiple daily injection treatment show the need for new treatments for this group of patients.

DETAILED DESCRIPTION:
This study evaluates between group change in glycemic control (HbA1c) after 6 months of insulin pump therapy in patients with type 2 Diabetes Mellitus, as compared to patients on multiple daily injections (MDI) therapy over the same time period. It also evaluates between group changes in diabetes clinical outcomes after 6 months in patients with type 2 DM. Patient related outcomes will be measured after 6 months of therapy. The primary endpoint will be between group difference in average HbA1c changes from baseline to 6 months, when comparing Continuous Subcutaneous Insulin Infusion (CSII) to MDI.

The secondary end point concerns the safety issues such as severe hypoglycemia incidence: defined as an episode absolutely requiring assistance from another person and preferably accompanied by a confirmatory blood glucose by finger stick of less than 50mg/dL (2.8 mmol/L), (i.e., subject is unable to treat self and requires carbohydrate, glucagon or other resuscitative actions to prevent further clinical deterioration), hospitalizations, Diabetic Ketoacidosis (DKA), an acute metabolic complication of diabetes, characterized by hyperglycemia, hyperketonemia, and metabolic acidosis, within group difference in HbA1c from 6 months to 12 months, change in weight or BMI, change in Lipids : total cholesterol, high density lipoprotein(HDL),low density lipoprotein(LDL),triglyceride, change in blood pressure, Insulin Dosage Changes (Total Daily Dose), Number of self monitoring blood glucose (SMBG)/day, treatment satisfaction: Diabetes Treatment Satisfaction Questionnaire status and change version (DTSQs and DTSQc).

The hypotheses underlying the secondary outcomes : the pump therapy improves glycaemic control whilst utilizing less total daily dose of insulin in comparison to multiple daily injections of insulin. This is associated with parallel improvement in metabolic profiles such as blood pressure and lipids. As for the glucose monitoring, investigators want to evaluate whether there is any difference in the frequency of SMBG/day between the 2 treatment groups. More frequent SMBG monitoring denotes better compliance, motivation and empowerment by the participants to control their diabetes.

ELIGIBILITY:
Inclusion Criteria:

CRITERIA FOR INCLUSION AT SCREENING

1. Diagnosed with type 2 Diabetes Mellitus, as per Investigator diagnosis
2. HbA1c (DCCT-standard) must be ≥ 9.0% and ≤12%
3. Insulin resistance defined as required daily dose up to 1.5u/kg or a maximum of 200 units insulin per day
4. Aged 20 to 75 years old inclusive
5. On premixed regimen (human or analogue insulin) defined as ≥ 2 injections per day for at least 3 months prior signing the informed consent
6. Ability to comply with technology, according to Investigator's judgment
7. Patients must be willing to undergo all study procedures
8. Female patients of child-bearing potential must be using adequate contraception means as assessed by Investigator

CRITERIA FOR INCLUSION AT RANDOMISATION

1. Diagnosed with type 2 DM, as per Investigator diagnosis
2. HbA1c (DCCT-standard) must be ≥ 9.0% and ≤12%
3. Insulin resistance defined as required daily dose up to 1.5 U/Kg or a maximum of 200 units per day
4. On premixed regimen (human or analogue insulin) defined as ≥ 2 injections per day for at least 3 months prior signing the informed consent
5. Ability to comply with technology, according to Investigator's judgment
6. ≥ 2.5 SMBG per day on average
7. Patients must be willing to undergo all study procedures
8. Female patients of child-bearing potential must be using adequate contraception means as assessed by Investigator

Exclusion Criteria:

CRITERIA FOR EXCLUSION (AT SCREENING AND RANDOMISATION)

1. Subject has a history (≥ 2 events) of hypoglycemic seizure or hypoglycemic coma within the last 6 months
2. Subject is pregnant as assessed by a pregnancy test with central laboratory, or plans to become pregnant during the course of the study
3. Participation in another interventional clinical study, on-going or completed less than 3 months prior to signature of Patient Informed Consent.
4. Subject has proliferative retinopathy or sight threatening maculopathy
5. Subject has

   * an acute coronary syndrome (myocardial infarction or unstable angina) within 12 months OR
   * coronary artery revascularization by bypass surgery or stenting within 3 months OR
   * a transient ischemic attack (TIA) or cerebrovascular accident (CVA) within 3 months OR
   * hospitalization for heart failure within 3 months or current New York Functional Class III or IV OR
   * current 2nd or 3rd degree heart block OR
   * symptomatic ventricular rhythm disturbances OR
   * thromboembolic disease within the last 3 months OR
6. Subject with renal impairment expressed as estimated glomerular filtration rate (eGFR) using the Modification of Diet in Renal Disease (MDRD) formula < 30 ml/min as demonstrated by the screening central laboratory value at the time of enrollment
7. Subject has taken oral or injectable steroids within the last 30 days.
8. Systolic blood pressure on screening visit is > 180 mmHg
9. Diastolic blood pressure on screening visit is > 110 mmHg
10. Any other disease (eg active cancer under treatment) or condition including abnormalities found on the screening tests, that in the opinion of the Investigator, may preclude the patient from participating in the study
11. Taking any medication prescribed for weight loss
12. Alcohol or drug abuse, other than nicotine, at the Investigator's discretion Use of a Glucagon Like Peptide-1 agonist or pramlintide (Symlin®). Glucagon Like Peptide-1 slows gastric emptying, thereby decreasing the rate of glucose absorption. Pramlintide (Symlin®) is a commercially available analogue of amylin, a synergistic partner to insulin.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
between group difference of HbA1c changes from baseline to 6 months | 6 months
  Between group difference in HbA1c changes from baseline to 6 months, when comparing CSII to MDI

SECONDARY OUTCOMES:
Within group difference in HbA1c changes from 6 months to 12 months | 1 year
  Within group difference in HbA1c changes from 6 months to 12 months after cross-over from MDI to CSII
Safety endpoints which are 1) Number of events of severe hypoglycemia 2)Any hospitalizations for hypoglycaemia or hyperglycaemic emergencies 3)Number of events of Diabetic Ketoacidosis (DKA) | 1 year
  1. Number of events of severe hypoglycemia : defined as an episode absolutely requiring assistance from another person and preferably accompanied by a confirmatory blood glucose by finger stick of less than 50mg/dL (2.8 mmol/L), (i.e., subject is unable to treat self and requires carbohydrate, glucagon or other resuscitative actions to prevent further clinical deterioration)
  2. Any hospitalizations for hypoglycaemia or hyperglycaemic emergencies
  3. Number of events of Diabetic Ketoacidosis (DKA), an acute metabolic complication of diabetes, characterized by hyperglycemia, hyperketonemia, and metabolic acidosis
change in weight (kg) | 1 year
  Between and within group difference in average weight changes when comparing CSII to MDI
Number of Self Monitoring Blood Glucose (SMBG) per day | 1 year
  Between and within group difference in the number of SMBG per day between CSII and MDI. The data is downloaded using Bayer Glucofacts Deluxe Software from the glucometer during each visit.
Total Daily Insulin Dosage per day in Unit/day | 1 year
  Between and within group total daily insulin dosage per day in Unit/day between CSII and MDI. The total daily insulin dose per day in the CSII group is downloaded from Medtronic CareLink Therapy Management Software whereas for the MDI group, it is the cumulative dosage of total insulin per day.
Total Daily Insulin Dosage per body weight in kilograms per day (Unit/kg/day) | 1 year
  Between and within group total daily insulin dosage per day (Outcome 6) divide by body weight in kilograms (Outcome 8) measured as (Unit/kg/day) for each patient,comparing between CSII and MDI
Body weight in kilograms | 1 year
  Between and within group body weight in kilograms, comparing between CSII and MDI
Treatment satisfaction using Diabetes Treatment Satisfaction Questionnaire DTSQs | 1 year
  Treatment satisfaction: Diabetes Treatment Satisfaction Questionnaire using DTSQs comparing between CSII and MDI

CONTACTS AND LOCATIONS:
Overall Officials: Noor Rafhati Adyani NR Abdullah, MBBS,MRCP, Principal Investigator — Putrajaya Hospital, Malaysia
Locations (1):
- Hospital Putrajaya, Putrajaya, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No